CLINICAL TRIAL: NCT02305667
Title: A Comparison of Three Videolaryngoscopes for Double-Lumen Tubes Intubation in Humans. A Randomized Controlled Study
Brief Title: Videolaryngoscopes for Double Lumen Tube Intubations
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Imam Abdulrahman Bin Faisal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Supportive Care
Other Study IDs: ANE-2014-11-27
Record Dates: First submitted 2014-11-27; First posted 2014-12-02 (Estimated); Last update posted 2017-01-24 (Estimated); Status verified 2017-01

CONDITIONS: Thoracic Surgery; Need for Double Lumen Tubes
Keywords: Laryngoscope; Macintosh; Glidescope®; King Vision™; Airtraq®; intubation; double lumen tube

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Macintosh (Placebo Comparator): Double lumen tube intubation using Macintosh laryngoscope
  Interventions: Device: Macintosh
- Glidescope® (Active Comparator): Double lumen tube intubation using Glidescope® videolaryngoscope
  Interventions: Device: Glidescope®
- Airtraq® (Active Comparator): Double lumen tube intubation using Airtraq® videolaryngoscope
  Interventions: Device: Airtraq®
- King Vision™ (Active Comparator): Double lumen tube intubation using King Vision™ videolaryngoscope
  Interventions: Device: King Vision™

INTERVENTIONS:
Device: Macintosh — double lumen tube intubation using the Macintosh laryngoscope
  Arms: Macintosh
Device: Glidescope® — double lumen tube intubation using the Glidescope® videolaryngoscope. The distal portion of a left-sided DLT will be angulated to the right concealing the distal orifice of the tracheal lumen. The DLT will be advanced directly through the vocal cords after initial 90° clockwise rotation, the stylet will be removed, and then the DLT will be advanced gently while rotating in a 180° couterclockwise direction
  Arms: Glidescope®
Device: Airtraq® — double lumen tube intubation using the Airtraq® videolaryngoscope.
  Arms: Airtraq®
Device: King Vision™ — double lumen tube intubation using the King Vision™ videolaryngoscope. the distal 21 cm of the left-sided DLT will be bended to replicate the curve of the non-channeled blade and the proximal curve of the DLT remains directed to the right side. Then, after initial 90° clockwise rotation, the bronchial cuff passes through the vocal cords, the stylet of the DLT will be withdrawn and the DLT will be rotated 180°counterclockwise while advancing the DLT to the desired depth.
  Arms: King Vision™

SUMMARY:
Introduction: Compared with the Macintosh laryngoscopy (MAC), the videolaryngoscopes (VL) provide superior glottis views and longer times to double-lumen tube (DLT) intubation. We hypothesize that the use of the King Vision™ (KVL) and the Airtraq® VLs may reduce the time for DLT intubation compared with the Glidescope® (GVL) and MAC in patients undergoing thoracic procedures.

Methods: One hundred-forty patients who will be scheduled for elective thoracic procedures using the DLT for one-lung ventilation will be randomly assigned to one of four groups (n=35 per group) to intubate using the MAC, GVL, Airtraq®, or KVL. Time to DLT intubation, glottis view, ease of intubation, number of optimization maneuvers, and failure to intubation (>150 s.) will be recorded.

DETAILED DESCRIPTION:
Several regional surveys among thoracic anesthesiologists showed that the double-lumen endobronchial tubes (DLT) is still the first choice for lung separation.[1-3] The introduction of videolaryngoscopes (VL) enables the use of the DLTs instead of a bronchial blockers for lung separation in patients with difficult airway.[4-5]

There are numerous VLs, including, stylets, channeled and traditional VLs. The GlideScope®-assisted DLT insertion (Verathon Inc., Bothell, WA, USA), has been associated with variable intubation durations according to the experience of the intubating operators, despite superior vocal cord views.[6-7] The channeled VL, like as the Airtraq® (Prodol Limited, Viscaya, Spain) and the standard non-channeled blade of the King Vision™ (KVL™) (King Systems, Indianapolis, IN, USA), may offer additional benefits for DLT intubation in patients with limited mouth opening or restricted neck movement, [8-10] in whom the use of traditional VL like as the Glidescope® could be difficult. This is because of the larger outer diameter, the distal curvature and the increased rigidity of the DLT.[11]

Of note, the longer intubation durations with the use of different VL-assisted DLT insertion could be shortened with building up the operator's experience.

Comparing the effects of the three studied VLs on the time to DLT intubation in humans has not yet been studied.

We hypothesize that time to successful DLT intubation using the channeled VL, namely, the Airtraq® and KVL™, will be shorter than with the Macintosh (MAC) laryngoscope and GlideScope® VL when used by non-expert anesthesiologists. We will compare the effects of the MAC, GlideScope®, Airtraq® and KVL™ on the time to DLT intubation, laryngoscopic view, ease of intubation, number of intubation attempts, and number of optimization maneuvers in patients undergoing thoracic procedures using DLTs for one-lung ventilation (OLV).

Standard monitoring, and bispectral index (BIS), or state and response entropy based depth of anesthesia, (GE Healthcare, Helsinki, Finland) will be applied to all patients. Neuromuscular blockade will be measured with a train of four stimulation (TOF) of the ulnar nerve. Invasive blood pressure monitoring will be achieved by cannulation of the radial artery. After preoxygenation, general anesthesia will be induced with propofol 1.5 to 3mg kg-1 and fentanyl 2-3 µg kg-1 or remifentanil 0.05-0.2 ug Kg-1 min-1, titrated to achieve a BIS value < 60 or a state entropy values of less than 50 and a difference between response and state entropy of less than 10. Rocuronium (0.6 mg kg-1) will be given to facilitate intubation with an appropriate sized left-sided DLT.

In all groups, during the insertion of the DLT, exercise caution to avoid damage to the tracheal cuff by the upper teeth during its passage through the mouth opening. After DLT intubation, the tracheal cuff will be inflated and ventilation of the lungs commenced. Then, the correct position of its tip will be confirmed with a fiberoptic bronchoscope.

The first intubation attempt will be considered a failure if the trachea is not successfully intubated within 150 s or if the peripheral oxygen saturation (SpO2) decreases by 5%. Following an initial tracheal intubation failure, the participants will be allowed to use any maneuver and device they would normally use to navigate the DLT into the trachea.

Demographic data will be recorded including grade, experience with the VLs, and previous DLT intubation experience with the VLs.

All data, with the exception of the difficulty of device use score, will be recorded by blinded investigators.

A pilot study showed that the mean time to DLT intubation using the GlideScope® VL was 72 seconds with a standard deviation of 45.2 seconds. An a priori power analysis indicated that a sample size of 32 participants was sufficiently large to detect a 50% difference in the time to DLT intubation, during the use of the channeled VL, a type-I error of 0.008 (0.05/6 possible comparisons) and a power of 90%. We will add more patients (10%) for a final sample size of 35 participants to compensate dropping out during the study.

Data will be tested for normality using Kolmogorov-Smirnov test. Categorical data will be analyzed using the Fisher's exact test. Repeated-measures analysis of variance (ANOVA) will be used for continuous parametric variables, and the differences will be corrected by the post hoc Bonferroni test. Kruskal-Wallis test will be used for nonparametric values, and post hoc pairwise comparisons will be performed using the Wilcoxon rank-sum t test Continuous data will be presented as mean (standard deviation, SD), ordinal data will be presented as median (inter-quartile range), and categorical data will be presented as number (%). A value of p< 0.05 will be considered to be statistically significant.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologists' physical status II/III
* Elective thoracic procedures

Exclusion Criteria:

* New York Heart Association (NYHA) functional classification class III to IV
* forced expiratory volume in 1 s (FEV1) less than 50% of predicted values
* forced vital capacity (FVC) less than 50% of predicted values
* severe asthma
* pregnancy
* risk of regurgitation
* risk of pulmonary aspiration
* history of gastro-esophageal reflux
* body mass index more than 40 kg m-2
* anticipated difficult intubation
* preoperative postoperative ventilatory support
* planned postoperative ventilatory support

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 133 (Actual)
Dates: Start 2015-05; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Time to the duration of endobronchial intubation | 3 minutes after laryngoscopy
  defined as the time from when the laryngoscope entered between the patient's lips until successful DLT placement (regardless of the number of attempts).[

SECONDARY OUTCOMES:
best obtained glottis view during laryngoscopy | 30 sec after laryngosocopy
  using Cormack and Lehane direct view or the 'video assisted view' seen on the video display screen
ease of endobronchial intubation | 30 sec after laryngosocopy
  a visual analogue score (VAS) of ease of endobronchial intubation (0 for much of ease and 100 for extremely difficult)
number of optimization maneuvers | 150 sec after laryngosocopy
number of the 'backwards upwards rightwards pressure' (BURP) maneuver | 150 sec after laryngosocopy
failure rate for double lumen tube intubation | 150 sec after laryngosocopy
sore throat | 48 hours after surgery
  throat using a VAS from 0, indicating 'none' to 10, 'severe' sore throat
hoarseness | 48 hours after surgery
  hoarseness using numerical scale observed by the anesthesiologist [0: absent, 1: subjective, or 3: aphonic]

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed R El Tahan, MD, Principal Investigator — Associate Professor at Anesthesiology Dept; Alaa khidr, MD, Study Director — Imam Abdulrahman Bin Faisal University
Locations (1):
- King Fahd Hospital of the University, Khobar, Eastern Province, Saudi Arabia